CLINICAL TRIAL: NCT06536725
Title: Observation of Clinical Consistency of Organoid-on-chips Drug Sensitivity Detection in Chemotherapy for Prostate Cancer Patients With Visceral Metastasis
Brief Title: Observation of Clinical Consistency of Organoid-chips Drug Sensitivity in Chemotherapy for PCa With Visceral Metastasis
Status: Recruiting | Type: Observational
Sponsor: Tianjin Medical University Second Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Organoid-on-chips-PCa
Record Dates: First submitted 2024-07-30; First posted 2024-08-05 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Prostate Cancer; Organoid
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — These samples are used for NGS detection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PCa Patients With Visceral Metastasis: Prostate cancer patients with visceral metastasis.
  Interventions: Other: Building Organoid-on-chips models

INTERVENTIONS:
Other: Building Organoid-on-chips models — This project obtains surgical or biopsy samples from prostate cancer patients with visceral metastasis for the construction of organoids.

SUMMARY:
This project plans to establish an organoid chip model of prostate cancer patients with internal organ metastasis from surgical or biopsy tissue sources, and test the sensitivity of commonly used chemotherapy drugs based on organoid chip drug sensitivity testing technology to screen out sensitive individualized treatment plans.

DETAILED DESCRIPTION:
This project plans to establish an organoid chip model of prostate cancer patients with internal organ metastasis from surgical or biopsy tissue sources, and test the sensitivity of commonly used chemotherapy drugs based on organoid chip drug sensitivity testing technology to screen out sensitive individualized treatment plans;The final medication regimen for patients is determined by doctors based on their experience and in vitro drug sensitivity results. The actual clinical efficacy of medication is tracked for patients, and the organoid chip drug sensitivity detection model is analyzed as a predictor of the sensitivity, specificity, and accuracy of anti-tumor chemotherapy drugs, providing data reference for clinical applications.At the same time, analyze the accuracy of drug sensitivity testing results and clinical empirical medication.If patients are treated with a chemotherapy combined with immunotherapy regimen, the in vitro sensitivity of immune drugs will be determined using organoid-immune co-culture technology, and exploratory research on the predictive performance of immune models will be conducted in conjunction with clinical medication.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with visceral metastasis of prostate cancer diagnosed clinically or pathologically;
2. Age ≥ 18 years old;
3. ECOG score ≤ 2 points or ECOG score 3-4 points due to tumor progression;
4. Normal liver and kidney function, serum transaminase ALT<66 U/L, AST<36 U/L, total bilirubin<22 umol/L, creatinine<106 umol/L, urea nitrogen<6.1 mmol/L; Normal bone marrow function: neutrophil count ≥ 1800/mm3 and platelet count ≥ 100000/mm3;
5. Can obtain surgical or biopsy samples;
6. Patients voluntarily join this study and sign an informed consent form.

Exclusion Criteria:

1. Patients with severe heart, liver, kidney, and peripheral nervous system diseases, as well as autoimmune diseases such as hyperthyroidism and hypothyroidism; Systemic lupus erythematosus, etc;
2. Patients who are unable to obtain tissue samples;
3. Subjects with active pulmonary tuberculosis (TB);
4. Subjects who are preparing for or have previously undergone tissue/organ transplantation;
5. Exclusion criteria are not listed, but the researchers believe that patients who are not suitable to participate in this clinical study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prostate Cancer Patients With Visceral Metastasis
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
ORR(Objective Response Rate) | 18 months
  Selecting ORR as the primary endpoint from clinical efficacy evaluation indicators.Evaluation of the best objective response rate (ORR) for each treatment according to RECIST 1.1. The best ORR is the best response reached during treatment according to RECIST 1.1 criteria.
Clinical Consistency | 18 months
  Sensitivity, specificity, and accuracy of drug sensitivity testing results based on successfully constructed organoids for predicting the main clinical efficacy evaluation indicators.

SECONDARY OUTCOMES:
Changes in tumor markers levels | 18 months
  The main tumor marker monitored is TPSA.The levels of PSA will be monitored every 3 (or 4) weeks for comparison to baseline levels until the time of PSA progression, as defined by PCWG3 criteria.The levels of other tumor markers will be monitored every 3 (or 4) weeks for comparison to baseline levels until the time of tumor markers progression.
PFS(Progression-free survival) | 18 months
  Progression-free survival (PFS) is defined as the time from the date of the first administration of patients medication plan based on organoids drug sensitivity test to the date of the first documentation of disease progression or death due to any cause, whichever comes first, censored at the last date at which the participant was determined to be progression-free.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical Unversity Second Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided